CLINICAL TRIAL: NCT03762408
Title: Comparative Study of the Efficacy and Safety of an Intra-articular Injection of ENKO 1 vs Durolane in Patients With Symptomatic Osteoarthritis of the Knee.
Brief Title: Efficacy and Safety of a Intra-articular Injection, ENKO1, in Patients With Symptomatic Knee Osteoarthritis.
Acronym: ENKORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Osteoarthritis Foundation International (OAFI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPK-ENK-2017-01
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Chondroitin Sulfate; Hyaluronic Acid; Intra-articular Injection; Viscosupplementation; Pain Relief; Biomarkers
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blinded (blind third party evaluation) The physician performing the infiltration will be different and cannot be related to the investigator evaluating the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENKO 1 (Experimental): ENKO 1 administered by single intra-articular injection.
  Interventions: Device: ENKO 1
- Durolane (Active Comparator): Durolane administered by single intra-articular injection.
  Interventions: Device: Durolane

INTERVENTIONS:
Device: ENKO 1 — 50 mg of HA/ 50 mg of CS in 5 ml
  Arms: ENKO 1
Device: Durolane — 60 mg HA crosslinked in 3 ml
  Arms: Durolane

SUMMARY:
Clinical trial with medical device, multicenter, single-blind (blind third party evaluation), randomized, comparative and in two paralell groups, to demonstrate the treatment according to usual clinical practice, of the combination of 50 mg Sodium Hyaluronate and 50 mg Chondroitin Sulfate (ENKO 1) in a single administration, has non-inferiority efficacy vs the comparator (Durolane; 60 mg HA crosslinked) in patients with symptomatic knee osteoarthritis after three months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Medial femorotibial compartment knee OA.
* Fulfilment of ACR criteria for knee OA (knee pain + grinding + stiffness in the morning < 30 minutes).
* Patients with a clinical course of disease longer than 6 months.
* Global pain score greater than 60 mm on a 0-100 mm VAS on the knee under study.
* Grade II or III according to the Kellgren and Lawrence classification system for the knee under study (on a posteroanterior X-ray performed under weight-bearing and for 6 months before randomisation).
* Patients taking analgesics for at least 3 months before randomisation and whom are dissatisfied with their current therapy.
* Patients who have given their consent in writing to take part in the study.
* Woman of childbearing age must take a urine pregnancy test which must be negative at the randomisation visit and be currently using an effective contraceptive method for at least 2 menstrual cycles (oral contraceptives, intrauterine device, tubal ligation or other effective procedures).

Exclusion Criteria:

* Isolated symptomatic patellofemoral osteoarthritis.
* Microcrystalline osteoarthritis.
* Prosthesis in knee under study.
* Joint lavage or arthroscopy or any surgery on the knee under study in the 6 months before randomisation.
* Paget's disease of bone, chondromatosis or villonodular sinovitis.
* Inflammatory, infectious or metabolic arthritis (rheumatoid arthritis, spondyloarthropathy or connective tissue diseases).
* Haemochromatosis, ochronosis or haemophilia.
* History of diseases that the investigator considers likely to interfere with the functional disability assessment.
* Knee surgery planned during the study period.

Other disease-related criteria:

* BMI greater than or equal to 30.
* Immunodeficiency or a serious or progressive disease (heart, lung, liver, kidney, haematological, neoplastic or infectious disease).
* Skin diseases or infections in the area of the injection site.
* Previous history of venous thromboembolism (including pulmonary embolism) or high risk of venous thromboembolism.
* Venous or lymphatic stasis of the leg under study.
* Severe acute or chronic disease that the investigator considers incompatible with the conduct of the study.
* Disease that the investigator considers likely to interfere with the study results or to expose the patient to an additional risk.
* Alcohol or drug abuse or dependence.

Previous or concomitant treatment-related criteria:

* Patients who have taken a SYSADOA, SERM or a drug/dietary supplement containing glucosamine, chondroitin sulfate, diacerein or avocado-soybean extracts in the 3 months before randomisation
* Patients who have taken paracetamol in the 24 hours before randomisation or any other symptomatic analgesic drug, including NSAIDs (except aspirin up to 325 mg/day for cardiovascular prophylaxis), in the 48 hours before randomisation
* Patients who have received any corticosteroid treatment by any route of administration (other than inhalers or the ocular or auricular routes) in the month before randomisation
* Patients who have received an intra-articular steroid injection in the knee under study in the month before randomisation or patients who have received intra-articular hyaluronic acid in the target knee in the 6 months before randomisation
* Patients who have received any local or topical treatment on the target knee in the 2 weeks before randomisation

Criteria related to concomitant medication:

* Hypersensitivity to paracetamol or NSAIDs

Study product-related criteria:

* Known allergy to the study treatments or to any of its ingredients.

Other criteria:

* Patients likely to be unable to comply with the protocol instructions and/or treatment, in the investigator's opinion
* Patients who have taken part in a clinical trial in the preceding 2 months or taking part in a trial at the time of randomisation
* Patients linguistically or mentally incapable of understanding the nature, objectives and possible consequences of the study; or who refuse to be subject to its limitations
* Patients who are family or colleagues (secretary, nurse, technician, etc.) of the investigator.
* Women: pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Pain Relief | Change from baseline pain relief at 6 months.
  Assessed using VAS (Visual Analogue Scale) Huskisson 0-100mm
  Pain relief scored on a scale of 0 to 10.
  0 means No pain and 10 means worst possible pain.

SECONDARY OUTCOMES:
Pain Relief | 0, 1, 6 and 12 weeks.
  Assessed using VAS (Visual Analogue Scale) Huskisson 0-100mm
  Pain relief scored on a scale of 0 to 10.
  0 means No pain and 10 means Worst possible pain.
Evaluation of functional WESTERN ONTARIO AND MCMASTER OSTEOARTHRITIS INDEX (WOMAC) index score (Pain subscale) | -7, 0, 1, 6, 12 and 24 weeks.
  Validated questionnaire for patients with osteoarthritis of the knee. 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Evaluation of functional WESTERN ONTARIO AND MCMASTER OSTEOARTHRITIS INDEX (WOMAC) index score (Stiffness subscale) | -7, 0, 1, 6, 12 and 24 weeks.
  Validated questionnaire for patients with osteoarthritis of the knee. 2 items: after first waking and later in the day. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Evaluation of functional WESTERN ONTARIO AND MCMASTER OSTEOARTHRITIS INDEX (WOMAC) index score (Functional capacity subscale) | -7, 0, 1, 6, 12 and 24 weeks.
  Validated questionnaire for patients with osteoarthritis of the knee. 17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Evaluation of percentage of patients who respond to treatment | 0, 1, 6, 12 and 24 weeks.
  Evaluation of percentage of patients who respond to treatment according to the OMERACT-OARSI criteria.
Global evaluation of the activity of the disease and of the respond to treatment by patient. | 0, 1, 6, 12 and 24 weeks.
  Global evaluation of the activity of disease by the patient (VAS (Visual Analogue Scale) from 0-100mm).
  Scale from 0 to 10, which correspond to: Mild (0-2), Moderate (3-7) and Intense (8-10).
  where 0 is better outcome and 10 is the worst outcome.
Evaluation of Health status of patients | 0, 1, 6, 12 and 24 weeks.
  Evaluation of Health status by quality of life questionnaire 12-Item Short Form Survey (SF-12).
  It consists of 12 items from the 8 dimensions of the SF-36 Physical Function, Social Function, Physical Role, Emotional Role, Mental Health, Vitality, Body Pain, General Health and evaluate intensity and frequency of each item.
  Scale ranges: Minimum 12 and maximum 60 scores. When 12 means better and 60 is the worse outcome.
Evaluation of concomitant medication intake | -7, 0, 1, 6, 12 and 24 weeks.
  Daily intake of Paracetamol (maximum 3g/day)
Evaluation of synovitis | -7, 0, 1, 6, 12 and 24 weeks.
  Clinical valoration of synovial joint swelling.
Biomarkers | -7 and 12 weeks
  Blood sample analysis of serum soluble biomarkers according to current validation by THE BIOMARKERS CONSORTIUM.
  Pre-selected biomarkers: Concentration of Serum CTXI, Serum NTXI, Serum-HA, Serum-PIIANP and Serum CTXII.
Adverse events | 0, 1, 6, 12 and 24 weeks.
  Number of Participants with any Adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Varela, Ph, MSc, Study Chair — OPKO Health, Inc.; Jordi Monfort, MD, PhD, Principal Investigator — Hospital del Mar
Locations (18):
- Spain (18):
  - Clínica Diagonal, Esplugues de Llobregat, Barceloma
  - Consell calatà de l'Esport, Esplugues de Llobregat, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Clínica Novo Sancti Petri, Chiclana de la Frontera, Cádiz
  - Clínica IQTRA, Torrejón de Ardoz, Madrid
  - Hospital de Torrelodones, Torrelodones, Madrid
  - Clínica Dr. Casermeiro, Mijas Costa, Málaga
  - Instituto Médico Arriaza, A Coruña
  - Hospital del Mar, Barcelona
  - Instituto POAL del Reumatología, Barcelona
  - Hospital Sant Rafael, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - BiClinic, Madrid
  - AMS Centro Médico del Ejercicio, Málaga
  - Clínica ISMEC, Seville
  - Clínica Gastaldi, Valencia
  - Clínica Traumatológica Dr. Baró, Valladolid
  - Hospital Vithas San José, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Undecided